CLINICAL TRIAL: NCT01233791
Title: Diazepam Vaginal Suppositories as a Treatment Option for High Tone PElvic Floor Dysfunction: A Randomized Controlled Trial.
Brief Title: Diazepam Vaginal Suppositories for High Tone Pelvic Floor Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10025-10-021
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Female Patients With High Tone Pelvic Floor Dysfunction
Keywords: high tone pelvic floor dysfunction; levator pain; dyspareunia
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal Diazepam Suppository (Experimental): Patients in this arm will be asked to use one vaginal suppository every night for 28 days
  Interventions: Drug: Vaginal Diazepam Suppository
- Vaginal Placebo Suppository (Placebo Comparator): Patients will be asked to use one vaginal suppository every night for 28 days
  Interventions: Drug: Placebo Suppository

INTERVENTIONS:
Drug: Vaginal Diazepam Suppository — 10mg compounded vaginal suppository
  Arms: Vaginal Diazepam Suppository
Drug: Placebo Suppository — Patients will be asked to use one vaginal suppository every night for 28 days
  Arms: Vaginal Placebo Suppository

SUMMARY:
The purpose of this study is to determine whether vaginal diazepam suppositories are an effective treatment of high tone pelvic floor dysfunction.

DETAILED DESCRIPTION:
High tone pelvic floor dysfunction is a common cause of pelvic pain in females. It is thought to be initiated by a sentinel event such as trauma, surgery, or vaginal delivery1. Currently, treatment options include warm baths, stretching, physical therapy with myofascial therapy or biofeedback, or pharmacologic therapy with oral amitriptyline or tiazadine2. Physical therapy can be effective. However, it usually involves frequent visits to a specialized physical therapist to undergo intravaginal treatments consisting of myofascial release, massage, or biofeedback. We would like to find a treatment option for patients that would be effective without the invasive and time consuming nature of physical therapy. It is known that diazepam is a valid treatment option for disorders involving spasticity including spastic cerebral palsy5 and tetanus. A literature search on diazepam and high tone pelvic floor dysfunction revealed one paper. This study has an intrinsic flaw as it is a retrospective chart review, and the results are confounded by concurrent physical therapy. They were, however, able to find that patients treated with diazepam suppositories showed a significant improvement in pelvic floor tone. They also assessed pain and sexual function, but these did not reach statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* candidates from the Division of Urogynecology at Good Samaritan Hospital in Cincinnati, OH
* aged 18-65
* high tone pelvic floor dysfunction

Exclusion Criteria:

* allergy to diazepam or any drug in the class of benzodiazepines
* current pelvic floor physical therapy
* pelvic surgery within the last 3 months
* current pregnancy, planning on pregnancy during the study period, or not sure if pregnant
* regular benzodiazepine, muscle relaxant, or daily alcohol use
* history of alcohol or drug abuse
* contraindications to diazepam: hepatic or renal dysfunction, myasthenia gravis, acute narrow angle glaucoma, severe respiratory insufficiency, sleep apnea

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Surface EMG | After 28 days of treatment
  A baseline sEMG will be compared to sEMG after 28 days of treatment.

SECONDARY OUTCOMES:
Surface EMG Midpoint | 14 days after treatment
  A baseline sEMG will be compared to sEMG after 14 days of treatment.
FSFI | 28 days
  Baseline FSFI scores will be compared to scores after 4 weeks of treatment to asses sexual function
VAS | 28 days
  Visual analog scale for pain will be collected at baseline and compared to VAS after 28 days of treatment
SF-12 | 28 days
  baseline SF-12 scores will be compared to SF-12 scores after 28 days of treatment to asses quality of life in the two domains of mental and physical well-being.
PGI-I | 28 days
  Patient Global Impression of Improvement will be asked after 28 days of treatment to determine if the patient felt the treatment was helpful
PGI-S | 28 days
  Patient Global Impression of Severity will be collected and compared to determine how severe teh patient perceived their condition to be before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Catrina C Crisp, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States